CLINICAL TRIAL: NCT03112603
Title: A Phase III Randomized Open-label Multi-center Study of Ruxolitinib vs. Best Available Therapy in Patients With Corticosteroid-refractory Chronic Graft vs Host Disease After Allogeneic Stem Cell Transplantation (REACH3)
Brief Title: A Study of Ruxolitinib vs Best Available Therapy (BAT) in Patients With Steroid-refractory Chronic Graft vs. Host Disease (GvHD) After Bone Marrow Transplantation (REACH3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-365 (REACH3); CINC424D2301 (Other: Novartis Pharmaceuticals); 2016-004432-38 (EudraCT Number)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2017-04-04; First posted 2017-04-13 (Actual); Results first posted 2022-04-15 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: Graft-versus-host disease (GvHD); Chronic GvHD (cGvHD); steroid-refractory; ruxolitinib; Janus kinase inhibitor
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — ruxolitinib; Photopheresis; Methotrexate; Mycophenolic Acid; Proto-Oncogene Proteins c-raf; Everolimus; Sirolimus; Infliximab; Rituximab; Pentostatin; Imatinib Mesylate; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): Ruxolitinib for the treatment period and extension period.
  Interventions: Drug: Ruxolitinib
- Best Available Therapy (Active Comparator): Best available therapy for the treatment period and extension period, with optional crossover to ruxolitinib after Cycle 6.
  Interventions: Drug: Extracorporeal photopheresis (ECP); Drug: Low-dose methotrexate (MTX); Drug: Mycophenolate mofetil (MMF); Drug: mechanistic Target of Rapamycin (mTOR) inhibitors (everolimus or sirolimus); Drug: Infliximab; Drug: Rituximab; Drug: Pentostatin; Drug: Imatinib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib twice daily at the protocol-defined starting dose.
  Other Names: Jakafi, INCB018424
  Arms: Ruxolitinib
Drug: Extracorporeal photopheresis (ECP) — Best available therapy (BAT) will be selected by the investigator for each participant. BAT may not include experimental agents (ie, those not approved for the treatment of any indication) as well as a limited number of other selected drugs in accordance with the protocol-defined requirements. The BAT in this study will be among the following treatments currently used in this setting (no other types or combinations of BATs are permitted in this study).
  Arms: Best Available Therapy
Drug: Low-dose methotrexate (MTX) — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: Mycophenolate mofetil (MMF) — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: mechanistic Target of Rapamycin (mTOR) inhibitors (everolimus or sirolimus) — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: Infliximab — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: Rituximab — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: Pentostatin — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: Imatinib — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy
Drug: Ibrutinib — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines for any dose adjustment.
  Arms: Best Available Therapy

SUMMARY:
The purpose of this study is to assess the efficacy of ruxolitinib against best available therapy in participants with steroid-refractory chronic graft-versus-host disease (SR cGvHD).

ELIGIBILITY:
Inclusion Criteria:

* Have undergone allogeneic stem cell transplantation (alloSCT) from any donor source (matched unrelated donor, sibling, haplo-identical) using bone marrow, peripheral blood stem cells, or cord blood. Recipients of non-myeloablative, myeloablative, and reduced intensity conditioning are eligible
* Evident myeloid and platelet engraftment: Absolute neutrophil count (ANC) > 1000/mm^3 and platelet count > 25,000/ mm^3
* Participants with clinically diagnosed moderate to severe cGvHD according to NIH Consensus Criteria prior to randomization:

  * Moderate cGvHD: At least one organ (not lung) with a score of 2, 3 or more organs involved with a score of 1 in each organ, or lung score of 1
  * Severe cGvHD: at least 1 organ with a score of 3, or lung score of 2 or 3
* Participants currently receiving systemic or topical corticosteroids for the treatment of cGvHD for a duration of < 12 months prior to Cycle 1 Day 1 (if applicable), and have a confirmed diagnosis of steroid-refractory cGvHD defined per 2014 NIH consensus criteria irrespective of the concomitant use of a calcineurin inhibitor (CNI), as follows:

  * A lack of response or disease progression after administration of minimum prednisone 1 mg/kg/day for at least 1 week, OR
  * Disease persistence without improvement despite continued treatment with prednisone at > 0.5 mg/kg/day or 1 mg/kg/every other day for at least 4 weeks, OR
  * Increase to prednisolone dose to > 0.25 mg/kg/day after 2 unsuccessful attempts to taper the dose
* Participant must accept to be treated with only one of the following BAT options on Cycle 1 Day 1 (additions and changes are allowed during the course of the study, but only with BAT from the following BAT options): extracorporeal photopheresis (ECP), low-dose methotrexate (MTX), mycophenolate mofetil (MMF), mTOR inhibitors (everolimus or sirolimus), infliximab, rituximab, pentostatin, imatinib, ibrutinib

Exclusion Criteria:

* Participants who have received 2 or more systemic treatment for cGvHD in addition to corticosteroids ± CNI for cGvHD
* Patients that transition from active aGvHD to cGvHD without tapering off corticosteroids ± CNI and any systemic treatment

  * Patients receiving up to 30 mg by mouth once a day of hydrocortisone (i.e., physiologic replacement dose) of corticosteroids are allowed.
* Participants who were treated with prior JAK inhibitors for aGvHD; except when the participant achieved complete or partial response and has been off JAK inhibitor treatment for at least 8 weeks prior to Cycle 1 Day 1
* Failed prior alloSCT within the past 6 months from Cycle 1 Day 1
* Participants with relapsed primary malignancy, or who have been treated for relapse after the alloSCT was performed
* Steroid refractory cGvHD occurring after a non-scheduled donor lymphocyte infusion (DLI) administered for preemptive treatment of malignancy recurrence. Participants who have received a scheduled DLI as part of their transplant procedure and not for management of malignancy relapse are eligible
* Any corticosteroid therapy for indications other than cGvHD at doses > 1 mg/kg/day methylprednisolone or equivalent within 7 days of Cycle 1 Day 1

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, Study Director — Incyte Corporation
Locations (170):
- United States (31):
  - Incyte Investigative Site, Tucson, Arizona
  - Incyte Investigative Site, Duarte, California
  - Incyte Investigative Site, La Jolla, California
  - Incyte Investigative Site, Los Angeles, California
  - Incyte Investigative Site, New Haven, Connecticut
  - Incyte Investigative Site, Wilmington, Delaware
  - Incyte Investigative Site, Gainesville, Florida
  - Incyte Investigative Site, Tampa, Florida
  - Incyte Investigative Site, Chicago, Illinois
  - Incyte Investigative Site, Maywood, Illinois
  - Incyte Investigative Site, Indianapolis, Indiana
  - Incyte Investigative Site, Westwood, Kansas
  - Incyte Investigative Site, Lexington, Kentucky
  - Incyte Investigative Site, Boston, Massachusetts
  - Incyte Investigative Site, Omaha, Nebraska
  - Incyte Investigative Site, Hackensack, New Jersey
  - Incyte Investigative Site, New York, New York
  - Incyte Investigative Site, Chapel Hill, North Carolina
  - Incyte Investigative Site, Durham, North Carolina
  - Incyte Investigative Site, Winston-Salem, North Carolina
  - Incyte Investigative Site, Cincinnati, Ohio
  - Incyte Investigative Site, Cleveland, Ohio
  - Incyte Investigative Site, Columbus, Ohio
  - Incyte Investigative Site, Oklahoma City, Oklahoma
  - Incyte Investigative Site, Philadelphia, Pennsylvania
  - Incyte Investigative Site, Pittsburgh, Pennsylvania
  - Incyte Investigative Site, Nashville, Tennessee
  - Incyte Investigative Site, Dallas, Texas
  - Incyte Investigative Site, Houston, Texas
  - Incyte Investigative Site, Seattle, Washington
  - Incyte Investigative Site, Milwaukee, Wisconsin
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Parkville, Victoria
- Austria (4):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (6):
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- Czechia (3):
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Hradec Králové, CZE
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense
- France (15):
  - Novartis Investigative Site, Bordeaux, Aquitaine
  - Novartis Investigative Site, Amiens Cedex1
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Benite Cédex
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (19):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Pátrai, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Novartis Investigative Site, Budapest, Hungary
- India (4):
  - Novartis Investigative Site, Navi Mumbai, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Delhi
  - Novartis Investigative Site, Vellore
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (15):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Perugia
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyō-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Okayama
- Novartis Investigative Site, Amman, Jordan
- Netherlands (4):
  - Novartis Investigative Site, Utrecht, The Netherlands
  - Novartis Investigative Site, Leiden
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Oslo, Norway
- Poland (5):
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Gliwice, Silesian Voivodeship
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigational Site, Lisbon
  - Novartis Investigative Site, Porto
- Incyte Investigative Site, Ponce, Puerto Rico
- Novartis Investigational Site, Bucharest, Romania
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Seoul, South Korea
- Spain (12):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, El Palmar, Murica
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Uppsala
- Switzerland (2):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeiser R, Russo D, Ram R, Hashmi SK, Chakraverty R, Middeke JM, Musso M, Giebel S, Uzay A, Langmuir P, Hamad N, Burock K, Gowda M, Stefanelli T, Lee SJ, Teshima T, Locatelli F. Ruxolitinib in Patients With Corticosteroid-Refractory or Corticosteroid-Dependent Chronic Graft-Versus-Host Disease: 3-Year Final Analysis of the Phase III REACH3 Study. J Clin Oncol. 2025 Aug 10;43(23):2566-2571. doi: 10.1200/JCO-24-02477. Epub 2025 Jun 25. PMID 40561385
- [Derived] Mahmoudjafari Z, Kintsch E, Xue Z, Bhatt V, Galvin J, Locatelli F, Zeiser R. Impact of concomitant azoles on ruxolitinib treatment in patients with GVHD: post hoc analyses of REACH2 and REACH3. Blood Adv. 2025 Aug 26;9(16):4206-4216. doi: 10.1182/bloodadvances.2025016212. PMID 40472328
- [Derived] Le RQ, Wang X, Zhang H, Li H, Przepiorka D, Vallejo J, Leong R, Ma L, Goldberg KB, Pazdur R, Theoret MR, De Claro A. FDA Approval Summary: Ruxolitinib for Treatment of Chronic Graft-Versus-Host Disease after Failure of One or Two Lines of Systemic Therapy. Oncologist. 2022 Jun 8;27(6):493-500. doi: 10.1093/oncolo/oyac042. PMID 35363318
- [Derived] Zeiser R, Polverelli N, Ram R, Hashmi SK, Chakraverty R, Middeke JM, Musso M, Giebel S, Uzay A, Langmuir P, Hollaender N, Gowda M, Stefanelli T, Lee SJ, Teshima T, Locatelli F; REACH3 Investigators. Ruxolitinib for Glucocorticoid-Refractory Chronic Graft-versus-Host Disease. N Engl J Med. 2021 Jul 15;385(3):228-238. doi: 10.1056/NEJMoa2033122. PMID 34260836
- [Derived] Jagasia M, Zeiser R, Arbushites M, Delaite P, Gadbaw B, Bubnoff NV. Ruxolitinib for the treatment of patients with steroid-refractory GVHD: an introduction to the REACH trials. Immunotherapy. 2018 Apr;10(5):391-402. doi: 10.2217/imt-2017-0156. Epub 2018 Jan 10. PMID 29316837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 29 countries globally. During the main treatment period, participants were randomly assigned to a ruxolitinib arm or a Best Available Therapy (BAT) arm for 6 cycles of treatment. At the end of Cycle 6, participants in the BAT arm either crossed over to ruxolitinib treatment or entered the survival follow-up phase.
Pre-assignment Details: A total of 404 participants were screened, of whom 72 were screen failures and 3 were not randomized for various reasons. Out of the 329 participants randomized, 6 did not receive BAT due to logistical reasons. A total of 329 participants were included in the Full Analysis Set (FAS); 165 were in the ruxolitinib arm and 164 were in the BAT arm.
Groups:
- Ruxolitinib: Ruxolitinib was administered orally twice per day at a dose of 10 milligrams (mg).
- Best Available Therapy: Participants received best available therapies (BATs), including, but not limited to, extracorporeal photopheresis (ECP), low-dose methotrexate (MTX), mycophenolate mofetil (MMF), mTOR inhibitors (everolimus or sirolimus), infliximab, rituximab, pentostatin, imatinib, and ibrutinib based on the investigator's decision.
- Ruxolitinib Cross-Over Period: Participants from the BAT arm at the end of Cycle 6 crossed over to ruxolitinib treatment.
Period: End of Randomization Period
Arm/Group | Ruxolitinib | Best Available Therapy | Ruxolitinib Cross-Over Period
Started | 165 | 164 | 0
Completed | 29 | 24 | 0
Not Completed | 136 | 140 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Participant/Guardian Decision | 7 | 14 | 0
Not completed — Physician Decision | 43 | 18 | 0
Not completed — Failure to Meet Protocol Continuation Criteria | 4 | 5 | 0
Not completed — Death | 10 | 7 | 0
Not completed — Disease Relapse | 12 | 7 | 0
Not completed — Lack of Efficacy | 25 | 77 | 0
Not completed — Adverse Event | 32 | 12 | 0
Period: End of Cross Over Period
Arm/Group | Ruxolitinib | Best Available Therapy | Ruxolitinib Cross-Over Period
Started | 0 | 0 | 70
Completed | 0 | 0 | 16
Not Completed | 0 | 0 | 54
Not completed — Death | 0 | 0 | 2
Not completed — Participant/Guardian Decision | 0 | 0 | 7
Not completed — Physician Decision | 0 | 0 | 29
Not completed — Lack of Efficacy | 0 | 0 | 8
Not completed — Adverse Event | 0 | 0 | 6
Not completed — Disease Relapse | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib | Best Available Therapy | Total
Number analyzed (Participants) | 165 | 164 | 329
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.9 (15.68) | 47.2 (16.17) | 46.5 (15.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 72 | 128
  Male | 109 | 92 | 201
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 116 | 132 | 248
  Black or African American | 2 | 0 | 2
  Asian | 33 | 21 | 54
  American Indian or Alaska Native | 2 | 0 | 2
  Other | 9 | 4 | 13
  Unknown | 3 | 7 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 13 | 13 | 26
  Not Hispanic/Latino | 118 | 115 | 233
  Not Reported | 26 | 25 | 51
  Unknown | 8 | 11 | 19
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Score has 6 grades (0-5). 0 = Fully active, able to carry out all pre-disease activities; 1 = Restricted in strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Active about 50% of waking hours; 3 = Capable of limited self-care, confined to bed/chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on self-care. Totally confined to bed/chair. 5 = Death.
  Participants
    0 | 39 | 42 | 81
    1 | 92 | 82 | 174
    2 | 22 | 22 | 44
    3 | 0 | 2 | 2
    Missing | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Ruxolitinib Versus Investigator's Choice Best Available Therapy (BAT) in Participants With Moderate or Severe Steroid Refractory Chronic Graft Versus Host Disease (SR-cGvHD) Assessed by Overall Response Rate (ORR) at the Cycle 7 Day 1 Visit
Description: ORR was defined as the percentage of participants in each arm demonstrating a complete response (CR) or partial response (PR) based on chronic GvHD (cGvHD) disease assessments (National Institutes of Health Consensus Criteria) without the requirement of additional systemic therapies for an earlier progression, mixed response, or non-response. Scoring of response was relative to the organ score at the time of randomization. CR: complete resolution of all signs and symptoms of cGVHD in all evaluable organs without the initiation or addition of new systemic therapy. PR: improvement in at least one organ (e.g., improvement of 1 or more points on a 4- to 7-point scale, or an improvement of 2 or more points on a 10- to 12-point scale) without progression in other organs or sites, initiation, or addition of new systemic therapies.
Time Frame: Cycle 7 Day 1 (each cycle was comprised of 4 weeks)
Population: Full Analysis Set (FAS): all participants to whom study treatment was assigned by randomization. Data reported are from the start of the study to Cycle 7 Day 1 (data cutoff of 08 May 2020).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
percentage of participants | 49.7 [41.8 to 57.6] | 25.6 [19.1 to 33.0]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.99, 95% CI 2-sided [1.86 to 4.80]

2. Secondary Outcome: Rate of Participants With Clinically Relevant Improvement of the Modified Lee cGvHD Symptom Scale Score
Description: To assess improvement of symptoms based on the total symptom score (TSS); a responder was defined as having achieved a clinically relevant reduction from Baseline of the TSS. The scale consists of 30 items in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological). Participants reported their level of symptom "bother" over the previous month on a 5-point likert scale: not at all, slightly, moderately, quite a bit, or extremely. Subscale scores and the summary score range from 0 to 100, with a higher score indicating worse symptoms.
Time Frame: Baseline; Cycle 7 Day 1 (each cycle was comprised of 4 weeks)
Population: FAS. Data reported are from the start of the study to Cycle 7 Day 1 (data cutoff of 08 May 2020).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
percentage of participants | 24.2 [17.9 to 31.5] | 11.0 [6.6 to 16.8]

3. Secondary Outcome: Rate of Failure-free Survival (FFS)
Description: Composite time to event endpoint incorporating the following FFS events: (i) relapse or recurrence of underlying disease or death due to underlying disease, (ii) nonrelapse mortality, or (iii) addition or initiation of another systemic therapy for cGvHD.
Time Frame: Baseline to when the last participant reached Cycle 7 Day 1 (each cycle was comprised of 4 weeks)
Population: FAS. Data reported are from the start of the study to Cycle 7 Day 1 (data cutoff of 08 May 2020).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
months | NA [18.6 to NA] — The median FFS time was not reached due to an insufficient number of participants with events. | 5.7 [5.6 to 6.5]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Other; p < 0.0001, Log Rank — The p-value was derived from a 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.370, 95% CI 2-sided [0.268 to 0.510] — The hazard ratio was obtained from a stratified Cox model using cGvHD severity at randomization as strata

4. Secondary Outcome: Rate of FFS at Study Completion
Description: as for outcome 3
Time Frame: From Baseline to Last Participant Last Visit (LPLV) (approximately 5 years)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
months | 38.4 [22.1 to NA] — The upper limit of the confidence interval was not estimable due to an insufficient number of participants with events. | 5.7 [5.6 to 6.5]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Other; Hazard Ratio (HR) = 0.361, 95% CI 2-sided [0.268 to 0.485] — The hazard ratio was obtained from a stratified Cox model using cGvHD severity at randomization as strata

5. Secondary Outcome: Best Overall Response (BOR) at Cycle 7 Day 1
Description: BOR was defined as the percentage of participants who achieved an overall response (CR+PR) based on cGvHD disease assessments (National Institutes of Health Consensus Criteria) without the requirement of additional systemic therapies for an earlier progression, mixed response, or non-response at any time point (up to Cycle 7 Day 1 or the start of additional systemic therapy for cGvHD). Scoring of response was relative to the organ score at the time of randomization. CR: complete resolution of all signs and symptoms of cGVHD in all evaluable organs without the initiation or addition of new systemic therapy. PR: improvement in at least one organ (e.g., improvement of 1 or more points on a 4- to 7-point scale, or an improvement of 2 or more points on a 10- to 12-point scale) without progression in other organs or sites, initiation, or addition of new systemic therapies. This analysis was based on the primary cutoff date (May 2020).
Time Frame: up to Cycle 7 Day 1 (each cycle was comprised of 4 weeks)
Population: FAS. Data reported are from the start of the study to Cycle 7 Day 1 (data cutoff of 08 May 2020).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
percentage of participants | 76.4 [69.1 to 82.6] | 60.4 [52.4 to 67.9]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Other; p = 0.0011, Cochran-Mantel-Haenszel — The one-sided p-value was calculated using a stratified Cochran-Mantel-Haenszel test; Odds Ratio (OR) = 2.17, 95% CI 2-sided [1.34 to 3.52] — The odds ratio and 95% confidence interval (CI) were calculated using a stratified Cochran-Mantel-Haenszel test

6. Secondary Outcome: BOR During Cross-over Treatment With Ruxolitinib
Description: BOR was defined as the percentage of participants who achieved an overall response (CR+PR) based on cGvHD disease assessments (National Institutes of Health Consensus Criteria) without the requirement of additional systemic therapies for an earlier progression, mixed response, or non-response at any time point (up to Cycle 7 Day 1 or the start of additional systemic therapy for cGvHD). Scoring of response was relative to the organ score at the time of randomization. CR: complete resolution of all signs and symptoms of cGVHD in all evaluable organs without the initiation or addition of new systemic therapy. PR: improvement in at least one organ (e.g., improvement of 1 or more points on a 4- to 7-point scale, or an improvement of 2 or more points on a 10- to 12-point scale) without progression in other organs or sites, initiation, or addition of new systemic therapies.
Time Frame: from Crossover Cycle 1 Day 1 to any time point up to and including Crossover Cycle 7 Day 1 (each cycle was comprised of 4 weeks)
Population: Cross-over Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Cross-Over Period
Number analyzed (Participants) | 70
percentage of participants | 81.4 [70.3 to 89.7]

7. Secondary Outcome: ORR at the End of Cycle 3
Description: ORR was defined as the percentage of participants in each arm demonstrating a CR or PR based on cGvHD disease assessments (National Institutes of Health Consensus Criteria) without the requirement of additional systemic therapies for an earlier progression, mixed response, or non-response. Scoring of response was relative to the organ score at the time of randomization. CR: complete resolution of all signs and symptoms of cGVHD in all evaluable organs without the initiation or addition of new systemic therapy. PR: improvement in at least one organ (e.g., improvement of 1 or more points on a 4- to 7-point scale, or an improvement of 2 or more points on a 10- to 12-point scale) without progression in other organs or sites, initiation, or addition of new systemic therapies.
Time Frame: Cycle 4 Day 1 (each cycle was comprised of 4 weeks)
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
percentage of participants | 54.5 [46.6 to 62.3] | 31.1 [24.1 to 38.8]
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — The one-sided p-value was calculated using a stratified Cochran-Mantel-Haenszel (CMH) test; Odds Ratio (OR) = 2.77, 95% CI 2-sided [1.75 to 4.39] — The odds ratio and 95% CI were calculated using a stratified CMH test

8. Secondary Outcome: Duration of Response Through Study Completion
Description: DOR was defined as the time from first response until cGvHD progression, death, or the date of change/addition of systemic therapies for cGvHD and as assessed for responders only. Response was based on cGvHD disease assessments (National Institutes of Health consensus criteria). Duration of response was evaluated in participants who achieved a CR or PR at or before Cycle 7 Day 1. The analysis included a larger number of participants than the number of participants who achieved CR or PR at Cycle 7 Day 1 (82 ruxolitinib and 42 BAT) because the analysis took into account not only those participants who achieved CR or PR at Cycle 7 Day 1, but also participants who achieved CR or PR before Cycle 7 Day 1 but who may have lost their response at Cycle 7 Day 1. For this reason, the number of participants in this analysis does not align with the best overall response (BOR) at Cycle 7 Day 1. This analysis was based on the cutoff date upon study completion (December 2022).
Time Frame: from first response to LPLV (approximately 5 years)
Population: FAS. Duration of response was evaluated in participants who achieved a CR or PR at or before Cycle 7 Day 1.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 126 | 103
Months | NA [NA to NA] — Median duration of response was not reached due to an insufficient number of participants with events. | 6.4 [4.9 to 11.4]

9. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: from the date of randomization to the date of death due to any cause up to LPLV (approximately 5 years)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
months | NA [NA to NA] — The median and upper and lower limits of the confidence interval were not estimable because too few participants died. | NA [41.0 to NA] — The median and upper limit of the confidence interval were not estimable because too few participants died.
Statistical Analysis 1: Comparison: Ruxolitinib vs Best Available Therapy; Test type: Other; p = 0.2396, Log Rank — The p-value was derived from a 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.851, 95% CI 2-sided [0.544 to 1.331] — The hazard ratio was obtained from a stratified Cox model using cGvHD severity at randomization as strata

10. Secondary Outcome: Cumulative Incidence of Non-relapse Mortality (NRM)
Description: Defined as the cumulative incidence rate from competing risk analysis for NRM from the date of randomization to the date of death not preceded by underlying disease relapse/recurrence.
Time Frame: Months 3, 6, 12, 18, 24, 30, and 36
Population: FAS. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
percentage of participants
  Month 3 | 5.45 [2.68 to 9.67] | 4.44 [1.96 to 8.48]
  Month 6: number analyzed (Participants) | 152 | 146
  Month 6 | 9.13 [5.34 to 14.15] | 6.43 [3.28 to 11.03]
  Month 12: number analyzed (Participants) | 143 | 137
  Month 12 | 15.30 [10.26 to 21.26] | 15.12 [9.94 to 21.30]
  Month 18: number analyzed (Participants) | 128 | 118
  Month 18 | 15.93 [10.78 to 21.98] | 16.48 [11.06 to 22.84]
  Month 24: number analyzed (Participants) | 121 | 114
  Month 24 | 17.83 [12.37 to 24.10] | 19.22 [13.36 to 25.90]
  Month 30: number analyzed (Participants) | 117 | 109
  Month 30 | 17.83 [12.37 to 24.10] | 19.22 [13.94 to 26.67]
  Month 36: number analyzed (Participants) | 114 | 106
  Month 36 | 17.83 [12.37 to 24.10] | 22.0 [15.73 to 28.96]

11. Secondary Outcome: Percentage of Participants With a ≥ 50% Reduction in Daily Corticosteroid Dose
Description: All corticosteroid dosages prescribed to the participant and all dose changes during the study were to be recorded for assessment of participants with a ≥ 50% reduction in daily corticosteroid dose.
Time Frame: from Day 15 up to Day 182
Population: Safety Set: all participants who received at least one dose of study treatment. Participants were to have been analyzed according to the study treatment received, where treatment received was defined as the randomized treatment if the participant took at least one dose of that treatment or the first treatment received if the randomized treatment was never received. Six participants in the BAT arm discontinued before receiving the first dose. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 158
percentage of participants
  Day 15 to ≤ Day 28: number analyzed (Participants) | 158 | 152
  Day 15 to ≤ Day 28 | 12.7 | 13.2
  Day 29 to ≤ Day 42: number analyzed (Participants) | 157 | 148
  Day 29 to ≤ Day 42 | 35.0 | 33.1
  Day 43 to ≤ Day 56: number analyzed (Participants) | 153 | 146
  Day 43 to ≤ Day 56 | 48.4 | 41.1
  Day 57 to ≤ Day 70: number analyzed (Participants) | 150 | 142
  Day 57 to ≤ Day 70 | 58.7 | 47.9
  Day 71 to ≤ Day 84: number analyzed (Participants) | 146 | 138
  Day 71 to ≤ Day 84 | 62.3 | 51.4
  Day 85 to ≤ Day 98: number analyzed (Participants) | 141 | 137
  Day 85 to ≤ Day 98 | 69.5 | 54.0
  Day 99 to ≤ Day 112: number analyzed (Participants) | 132 | 134
  Day 99 to ≤ Day 112 | 71.2 | 60.4
  Day 113 to ≤ Day 126: number analyzed (Participants) | 127 | 130
  Day 113 to ≤ Day 126 | 73.2 | 66.2
  Day 127 to ≤ Day 140: number analyzed (Participants) | 125 | 123
  Day 127 to ≤ Day 140 | 72.8 | 68.3
  Day 141 to ≤ Day 154: number analyzed (Participants) | 120 | 120
  Day 141 to ≤ Day 154 | 70.0 | 68.3
  Day 155 to ≤ Day 168: number analyzed (Participants) | 118 | 116
  Day 155 to ≤ Day 168 | 74.6 | 71.6
  Day 169 to ≤ Day 182: number analyzed (Participants) | 116 | 89
  Day 169 to ≤ Day 182 | 81.9 | 88.8

12. Secondary Outcome: Percentage of Participants Successfully Tapered Off of All Corticosteroids
Description: All corticosteroid dosages prescribed to the participant and all dose changes during the study were to be recorded for assessment of participants who successfully tapered off of all corticosteroids. Participants who completely tapered off corticosteroids refer to those who permanently discontinued steroids as per the dose administration panel and who did not restart steroids in the same interval. Participants who were tapered off and continued follow-up were also counted as being tapered off with 0 dose in subsequent intervals until they discontinued from the main treatment period or restarted steroid treatment.
Time Frame: up to Day 179
Population: FAS. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 158
percentage of participants
  Day 1 to ≤ Day 28 | 2.5 | 2.6
  Day 29 to ≤ Day 56 | 9.6 | 5.4
  Day 57 to ≤ Day 84 | 14.0 | 8.5
  Day 85 to ≤ Day 112 | 16.3 | 10.3
  Day 113 to ≤ Day 140 | 19.7 | 12.4
  Day 141 to ≤ Day 168 | 24.2 | 16.8
  Day 169 to ≤ Day 179 | 24.1 | 15.9

13. Secondary Outcome: Cumulative Incidence of Malignancy Relapse/Recurrence (MR)
Description: Defined as the cumulative incidence rate from competing risk analysis of MR from the date of randomization to hematologic malignancy relapse/recurrence.
Time Frame: Months 3, 6, 12, 18, 24, 30, and 36
Population: FAS. Cumulative incidence was calculated for participants with underlying hematologic malignant disease. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 156 | 160
percentage of participants
  0 to < 3 months | 1.92 [0.52 to 5.12] | 1.31 [0.26 to 4.27]
  3 to < 6 months: number analyzed (Participants) | 143 | 142
  3 to < 6 months | 3.22 [1.20 to 6.93] | 2.65 [0.87 to 6.21]
  6 to < 12 months: number analyzed (Participants) | 134 | 133
  6 to < 12 months | 5.18 [2.42 to 9.49] | 6.08 [2.98 to 10.73]
  12 to < 18 months: number analyzed (Participants) | 121 | 114
  12 to < 18 months | 7.82 [4.25 to 12.77] | 6.08 [2.98 to 10.73]
  18 to < 24 months: number analyzed (Participants) | 115 | 110
  18 to < 24 months | 8.48 [4.74 to 13.57] | 6.08 [2.98 to 10.73]
  24 to <30 months: number analyzed (Participants) | 111 | 105
  24 to <30 months | 8.48 [4.74 to 13.57] | 6.78 [3.46 to 11.62]
  30 to <36 months: number analyzed (Participants) | 108 | 102
  30 to <36 months | 8.48 [4.74 to 13.57] | 7.50 [3.96 to 12.52]

14. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT)
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The FACT-BMT is a 50-item self-report questionnaire that measures the effect of a therapy on domains including physical, functional, social/family, and emotional well-being, together with additional concerns relevant for bone marrow transplantation participants. The questions were based on a 5-point Likert scale, where 0 corresponds to "not at all" and 4 corresponds to "very much." The higher the final score, the better the quality of life. The FACT-BMT total score ranges from 0 to 148.
Time Frame: Baseline; up to Cycle 39 Day 1 (each cycle was comprised of 4 weeks)
Population: FAS. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
scores on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 122 | 102
  Cycle 2 Day 1 | 2.32 (12.191) | -0.22 (14.949)
  Cycle 3 Day 1: number analyzed (Participants) | 115 | 106
  Cycle 3 Day 1 | 0.62 (14.452) | -1.82 (15.849)
  Cycle 4 Day 1: number analyzed (Participants) | 110 | 100
  Cycle 4 Day 1 | 1.98 (15.888) | -1.05 (16.147)
  Cycle 5 Day 1: number analyzed (Participants) | 107 | 91
  Cycle 5 Day 1 | 1.25 (14.577) | -0.23 (18.903)
  Cycle 6 Day 1: number analyzed (Participants) | 96 | 85
  Cycle 6 Day 1 | 2.91 (14.562) | 2.41 (14.766)
  Cycle 7 Day 1: number analyzed (Participants) | 90 | 88
  Cycle 7 Day 1 | 4.14 (14.669) | 0.85 (16.811)
  Cycle 9 Day 1: number analyzed (Participants) | 88 | 46
  Cycle 9 Day 1 | 5.32 (16.815) | 1.20 (17.635)
  Cycle 12 Day 1: number analyzed (Participants) | 68 | 35
  Cycle 12 Day 1 | 7.26 (19.296) | 3.74 (18.059)
  Cycle 15 Day 1: number analyzed (Participants) | 59 | 31
  Cycle 15 Day 1 | 5.07 (18.220) | 7.58 (17.063)
  Cycle 18 Day 1: number analyzed (Participants) | 55 | 27
  Cycle 18 Day 1 | 4.10 (19.440) | 8.19 (17.993)
  Cycle 21 Day 1: number analyzed (Participants) | 56 | 24
  Cycle 21 Day 1 | 5.24 (19.485) | 3.68 (17.378)
  Cycle 24 Day 1: number analyzed (Participants) | 50 | 23
  Cycle 24 Day 1 | 5.90 (19.662) | 7.84 (18.561)
  Cycle 27 Day 1: number analyzed (Participants) | 50 | 21
  Cycle 27 Day 1 | 6.23 (18.880) | 5.10 (18.885)
  Cycle 30 Day 1: number analyzed (Participants) | 48 | 19
  Cycle 30 Day 1 | 7.53 (20.314) | 5.75 (21.037)
  Cycle 33 Day 1: number analyzed (Participants) | 49 | 19
  Cycle 33 Day 1 | 5.17 (20.330) | 5.67 (22.573)
  Cycle 36 Day 1: number analyzed (Participants) | 47 | 18
  Cycle 36 Day 1 | 8.72 (18.710) | 4.77 (24.186)
  Cycle 39 Day 1: number analyzed (Participants) | 50 | 18
  Cycle 39 Day 1 | 8.65 (21.669) | 6.64 (22.384)

15. Secondary Outcome: Change From Baseline in EQ-5D-5L
Description: The EQ-5D-5L is a descriptive classification consisting of five dimensions of health: mobility, self-care, usual activities, anxiety/depression, and pain/discomfort. The five-level version (no problems, slight problems, moderate problems, severe problems, and extreme problems) uses a 5-point Likert scale, with 1 being no problems and 5 being extreme problems.
Time Frame: Baseline; up to Cycle 39 Day 1 (each cycle was comprised of 4 weeks)
Population: FAS. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 164
scores on a scale
  Cycle 2 Day 1: number analyzed (Participants) | 118 | 98
  Cycle 2 Day 1 | 0.03 (0.214) | -0.01 (0.163)
  Cycle 3 Day 1: number analyzed (Participants) | 113 | 103
  Cycle 3 Day 1 | 0.03 (0.221) | -0.04 (0.259)
  Cycle 4 Day 1: number analyzed (Participants) | 108 | 97
  Cycle 4 Day 1 | 0.04 (0.196) | -0.01 (0.192)
  Cycle 5 Day 1: number analyzed (Participants) | 105 | 88
  Cycle 5 Day 1 | 0.02 (0.210) | -0.03 (0.243)
  Cycle 6 Day 1: number analyzed (Participants) | 96 | 81
  Cycle 6 Day 1 | 0.05 (0.230) | 0.01 (0.186)
  Cycle 7 Day 1: number analyzed (Participants) | 89 | 86
  Cycle 7 Day 1 | 0.07 (0.234) | -0.00 (0.225)
  Cycle 9 Day 1: number analyzed (Participants) | 86 | 42
  Cycle 9 Day 1 | 0.07 (0.228) | -0.02 (0.166)
  Cycle 12 Day 1: number analyzed (Participants) | 68 | 34
  Cycle 12 Day 1 | 0.07 (0.187) | 0.02 (0.158)
  Cycle 15 Day 1: number analyzed (Participants) | 60 | 30
  Cycle 15 Day 1 | 0.07 (0.250) | 0.03 (0.140)
  Cycle 18 Day 1: number analyzed (Participants) | 56 | 25
  Cycle 18 Day 1 | 0.07 (0.299) | 0.02 (0.110)
  Cycle 21 Day 1: number analyzed (Participants) | 57 | 24
  Cycle 21 Day 1 | 0.08 (0.268) | -0.00 (0.222)
  Cycle 24 Day 1: number analyzed (Participants) | 51 | 22
  Cycle 24 Day 1 | 0.07 (0.272) | 0.01 (0.164)
  Cycle 27 Day 1: number analyzed (Participants) | 49 | 21
  Cycle 27 Day 1 | 0.06 (0.299) | 0.03 (0.182)
  Cycle 30 Day 1: number analyzed (Participants) | 48 | 19
  Cycle 30 Day 1 | 0.05 (0.261) | 0.01 (0.159)
  Cycle 33 Day 1: number analyzed (Participants) | 50 | 19
  Cycle 33 Day 1 | 0.00 (0.282) | 0.05 (0.186)
  Cycle 36 Day 1: number analyzed (Participants) | 47 | 18
  Cycle 36 Day 1 | 0.06 (0.231) | 0.04 (0.216)
  Cycle 39 Day 1: number analyzed (Participants) | 50 | 18
  Cycle 39 Day 1 | 0.06 (0.255) | 0.01 (0.214)

16. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: Adverse events were defined as the appearance of (or worsening of any pre-existing) undesirable signs, symptoms, or medical conditions that occurred after the participant's signed informed consent was obtained. Abnormal laboratory values or test results occurring after informed consent constituted adverse events only if they induced clinical signs or symptoms, were considered clinically significant, required therapy (e.g., hematologic abnormality that required transfusion or hematological stem cell support), or required changes in study medication(s). TEAEs were defined as those AEs that started or worsened during the on-treatment period (either randomized or cross-over period).
Time Frame: from Baseline to LPLV (approximately 5 years)
Population: Safety Set. Six participants in the BAT arm discontinued before receiving the first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib | Best Available Therapy | Ruxolitinib Cross-Over Period
Number analyzed (Participants) | 165 | 158 | 70
Participants | 165 | 148 | 70

17. Secondary Outcome: Cmax of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: Cmax was defined as the maximum observed plasma concentration of ruxolitinib. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: Extensive Sampling Schedule: Cycle 1 Days 1 and 15: predose; 0.5, 1, 1.5, 4, 6, and 9 hours post-dose. Sparse Sampling Schedule: Cycle 1 Days 1 and 15: predose; 1.5 hours post-dose
Population: Pharmacokinetic Analysis Set (PAS): all participants who provided at least one evaluable pharmacokinetic (PK) concentration. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 20
nanograms per milliliter (ng/mL)
  Day 1 | 167 (39.3)
  Day 15: number analyzed (Participants) | 16
  Day 15 | 215 (48.8)

18. Secondary Outcome: AUClast of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: AUClast was defined as the area under the concentration-time curve up to the last measurable concentration of ruxolitinib. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: as for outcome 17
Population: PAS. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 20
ng*hour/mL
  Day 1 | 636 (40.8)
  Day 15: number analyzed (Participants) | 16
  Day 15 | 945 (56.1)

19. Secondary Outcome: AUCinf of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: AUCinf was defined as the area under the concentration-time curve from time 0 to infinity. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: as for outcome 17
Population: PAS. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hour/mL
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 10
ng*hour/mL
  Day 1 | 642 (32.7)
  Day 15: number analyzed (Participants) | 0

20. Secondary Outcome: CL/F of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: CL/F was defined as the oral dose clearance of ruxolitinib. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: as for outcome 17
Population: PAS. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 20
Liters/hour
  Day 1: number analyzed (Participants) | 10
  Day 1 | 15.6 (32.7)
  Day 15: number analyzed (Participants) | 7
  Day 15 | 15.2 (20.4)

21. Secondary Outcome: Vz/F of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: Vz/F was defined as the apparent oral dose volume of distribution of ruxolitinib. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: as for outcome 17
Population: PAS. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 20
Liters
  Day 1: number analyzed (Participants) | 10
  Day 1 | 54.0 (25.0)
  Day 15: number analyzed (Participants) | 7
  Day 15 | 50.9 (33.9)

22. Secondary Outcome: Tmax of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: tmax was defined as the time to reach the maximum plasma concentration of ruxolitinib. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: as for outcome 17
Population: PAS. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 20
hours
  Day 1 | 0.833 [0.417 to 4.08]
  Day 15: number analyzed (Participants) | 16
  Day 15 | 1.00 [0.417 to 2.00]

23. Secondary Outcome: t1/2 of Ruxolitinib After Single (Cycle 1 Day 1) and Multiple (Cycle 1 Day 15) Doses
Description: t1/2 was defined as the apparent terminal phase disposition half-life of ruxolitinib. Early enrolling participants (approximately the first 8 adult and first 4 adolescent participants) randomized to ruxolitinib arm followed an "extensive PK" sampling schedule. Subsequent participants randomized to ruxolitinib, any randomized participants receiving ruxolitinib after Cycle 6, and any randomized participants receiving BAT that cross over to ruxolitinib followed the "sparse PK" sampling schedule.
Time Frame: as for outcome 17
Population: PAS. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 20
hours
  Day 1: number analyzed (Participants) | 10
  Day 1 | 2.40 (28.9)
  Day 15: number analyzed (Participants) | 7
  Day 15 | 2.32 (19.8)

24. Secondary Outcome: Utilization of Medical Resources
Description: The percentage of participants with at least one submission to healthcare encounter was assessed.
Time Frame: from Baseline to LPLV (approximately 5 years)
Population: Safety Set. Six participants in the BAT arm discontinued before receiving the first dose.
Measure: Number; unit: percentage of participants
Arm/Group | Ruxolitinib | Best Available Therapy
Number analyzed (Participants) | 165 | 158
percentage of participants | 57.0 | 65.8

ADVERSE EVENTS:
Time Frame: from Baseline to LPLV (approximately 5 years)
Description: Treatment-emergent adverse events, defined as adverse events that started or worsened during the on-treatment period (either Randomized or Cross-over Period), have been reported for the Safety Set, which included participants who received at least one dose of drug. A total of 6 participants in the BAT arm discontinued before receiving the first dose.
Arm/Group | Ruxolitinib | Best Available Therapy | Ruxolitinib Cross-Over Period
All-Cause Mortality (participants affected / at risk) | 37/165 | 40/158 | 10/70
Serious Adverse Events (participants affected / at risk) | 86/165 | 71/158 | 27/70
Other Adverse Events (participants affected / at risk) | 158/165 | 132/158 | 62/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=165) | Best Available Therapy (N=158) | Ruxolitinib Cross-Over Period (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Spleen disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0
Corneal erosion (Eye disorders) | 1 | 0 | 0
Corneal perforation (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1
General physical health deterioration (General disorders) | 1 | 2 | 0
Generalised oedema (General disorders) | 1 | 1 | 0
Hyperthermia (General disorders) | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Necrosis (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 11 | 7 | 3
Stenosis (General disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Abdominal wall infection (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
Adenovirus reactivation (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Bacterial translocation (Infections and infestations) | 1 | 0 | 0
Brain abscess (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 3 | 4 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 3 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | 1 | 0
Dacryocanaliculitis (Infections and infestations) | 0 | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 2 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 4 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 1
Large intestine infection (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 1 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0
Measles (Infections and infestations) | 1 | 0 | 0
Meningitis cryptococcal (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumococcal infection (Infections and infestations) | 1 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 24 | 18 | 5
Pneumonia bacterial (Infections and infestations) | 3 | 2 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 2 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 1 | 0
Pulmonary nocardiosis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 3
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 4 | 1 | 1
Septic shock (Infections and infestations) | 2 | 4 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0
Systemic infection (Infections and infestations) | 1 | 1 | 0
Systemic mycosis (Infections and infestations) | 0 | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 1 | 0
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Alveolar proteinosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Loss of personal independence in daily activities (Social circumstances) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=165) | Best Available Therapy (N=158) | Ruxolitinib Cross-Over Period (N=70)
Anaemia (Blood and lymphatic system disorders) | 56 | 25 | 15
Leukopenia (Blood and lymphatic system disorders) | 10 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 25 | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 14 | 7
Cataract (Eye disorders) | 4 | 6 | 5
Dry eye (Eye disorders) | 11 | 10 | 2
Abdominal pain (Gastrointestinal disorders) | 7 | 9 | 4
Constipation (Gastrointestinal disorders) | 14 | 10 | 5
Diarrhoea (Gastrointestinal disorders) | 27 | 23 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 4
Nausea (Gastrointestinal disorders) | 19 | 21 | 3
Vomiting (Gastrointestinal disorders) | 15 | 12 | 3
Asthenia (General disorders) | 4 | 4 | 5
Fatigue (General disorders) | 25 | 15 | 7
Oedema peripheral (General disorders) | 13 | 18 | 4
Pyrexia (General disorders) | 34 | 16 | 9
BK virus infection (Infections and infestations) | 9 | 2 | 3
Bronchitis (Infections and infestations) | 7 | 3 | 7
COVID-19 (Infections and infestations) | 8 | 1 | 5
Conjunctivitis (Infections and infestations) | 13 | 6 | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 8 | 15 | 4
Influenza (Infections and infestations) | 16 | 10 | 2
Nasopharyngitis (Infections and infestations) | 17 | 10 | 1
Pneumonia (Infections and infestations) | 8 | 11 | 6
Upper respiratory tract infection (Infections and infestations) | 19 | 15 | 12
Urinary tract infection (Infections and infestations) | 13 | 9 | 4
Alanine aminotransferase increased (Investigations) | 32 | 8 | 5
Amylase increased (Investigations) | 12 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 19 | 6 | 3
Blood alkaline phosphatase increased (Investigations) | 12 | 6 | 3
Blood cholesterol increased (Investigations) | 15 | 7 | 1
Blood creatine phosphokinase increased (Investigations) | 11 | 1 | 2
Blood creatinine increased (Investigations) | 29 | 8 | 4
Fibrin D dimer increased (Investigations) | 9 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 19 | 7 | 3
Lipase increased (Investigations) | 10 | 4 | 3
Platelet count decreased (Investigations) | 19 | 11 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 2 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 6 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 4 | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16 | 14 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 9 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 22 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 11 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 13 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 10 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 7 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 5 | 1
Headache (Nervous system disorders) | 17 | 14 | 6
Tremor (Nervous system disorders) | 7 | 8 | 0
Insomnia (Psychiatric disorders) | 13 | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 15 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 10 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8 | 1
Hypertension (Vascular disorders) | 33 | 21 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03112603/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT03112603/SAP_001.pdf